CLINICAL TRIAL: NCT00318591
Title: A Prospective, Randomized, Parallel-group, Multi-center Study to Compare the Occurrence of Urinary Tract Infections in Patients With Spinal Cord Injury Using Either Coated or Uncoated Intermittent Catheters.
Brief Title: Comparative Study of Intermittent Catheters and Occurrence of Urinary Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DK046CC
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Results first posted 2011-05-25 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2015-08

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SpeediCath (Experimental): hydrophilic-coated intermittent catheter
  Interventions: Device: SpeediCath
- Conveen Uncoated (Experimental): uncoated urinary intermittent catheter
  Interventions: Device: Conveen Uncoated

INTERVENTIONS:
Device: SpeediCath — hydrophilic coated urinary intermittent catheter
  Other Names: Coated Catheter
  Arms: SpeediCath
Device: Conveen Uncoated — Uncoated urinary intermittent catheter
  Other Names: Uncoated catheter
  Arms: Conveen Uncoated

SUMMARY:
The purpose of this study is to investigate the frequency of urinary tract infections with symptoms in spinal cord injured patients requiring intermittent catheterization for emptying the bladder. Patients will use either a coated catheter or an uncoated catheter with gel.

DETAILED DESCRIPTION:
Introduction:

Spinal cord injured (SCI) constitutes a large group of patients suffering from neurogenic bladder dysfunction, which is often managed by intermittent catheterization (IC). Intermittent catheterization is accepted as a safe and effective method for maintaining bladder and renal health in individuals with neurogenic bladder dysfunction. However, IC several times a day places an individual at risk for urethral trauma, hematuria, and particularly symptomatic urinary tract infections (UTI).

Attempts to control UTI with prophylactic antibiotics or sterile technique have not been overly successful but more recent advances in catheter technology, such as the hydrophilic-coated catheter, offer potential benefit. The hydrophilic-coated catheter has a slippery, pre-lubricated surface (along the entire length of the catheter) when soaked in water, allowing smooth insertion without the need for additional water soluble lubricant. Two proposed advantages over uncoated catheters are 1) reduced incidence of symptomatic UTI, and 2) reduction of urethral irritation or urethral trauma, and lowered risk of urethral strictures. Currently, while there are trends in favour of hydrophilic-coated catheters with respect to UTI overall evidence remains inadequate for clinical decision-making for choice of catheter type. Randomised trials to date have been limited by short follow up, heterogeneity, attrition, imprecise outcome measures, and varying definitions of UTI5. Conclusions of the Cochrane group in 20076 were echoed in a recent comprehensive re-view of all studies on hydrophilic-coated catheters - there is modest evidence favouring hydrophilic-coated catheter in reduction of UTI, but further robust research is required.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic spinal cord injury within 3 months prior to inclusion
* Neurogenic bladder dysfunction requiring intermittent catheterization at least 3 times daily

Exclusion Criteria:

* Has symptoms of UTI at inclusion
* Treated with prophylactic antibiotics to prevent UTIs
* Has a history of unresolved bladder-ureteral reflux and/or stones in the urinary tract
* Has used intermittent catheterization for more than 10 days prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2006-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Cardenas, MD, Principal Investigator — University of Miami
Locations (16):
- United States (12):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Craig Hospital, Englewood, Colorado
  - University of Miami, Miami, Florida
  - Shepherd Center, Atlanta, Georgia
  - Boston Medical School, Boston, Massachusetts
  - University of Michigan Helaths Systems, Ann Arbor, Michigan
  - Mayo Clinic, Saint Mary Hospital MB3CF Rehabilitation, Rochester, Minnesota
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - The Institute for Rehabilitation and Research (TIRR), Houston, Texas
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - G.F.Strong Rehabilitation Centre, Vancouver, British Columbia
  - Parkwood Rehabilitation Centre, London, Ontario
  - Toronto Rehabilitation Centre, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- SpeediCath: Hydrophilic coated intermittent catheter
- Conveen Uncoated: Uncoated intermittent catheter
Period: Overall Study
Arm/Group | SpeediCath | Conveen Uncoated
Started | 105 | 114
Completed | 45 | 69
Not Completed | 60 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SpeediCath | Conveen Uncoated | Total
Number analyzed (Participants) | 105 | 114 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (14.4) | 35.1 (13.2) | 36.1 (13.8)
Sex/Gender, Customized [Number; unit: participants] — Gender is unknown for one participant
  participants
    Female | 22 | 20 | 42
    Male | 83 | 93 | 176
Region of Enrollment [Number; unit: participants]
  United States | 80 | 86 | 166
  Canada | 25 | 28 | 53

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Symptomatic Urinary Tract Infections (UTIs)
Description: Occurrence of symptomatic urinary tract infections (UTIs). Time to first UTI
Time Frame: 4-6 months
Population: ITT-population, symptomatic urinary tract infections treated with antibiotics
Measure: Number; unit: participants
Groups:
- SpeediCath Catheter: Hydrophilic coated intermittent catheter
Arm/Group | SpeediCath Catheter | Conveen Uncoated
Number analyzed (Participants) | 105 | 114
participants
  Free of UTIs from study start to day 30 | 19 (0) | 20 (0)
  Free of UTIs from study start to day 150 | 2 | 0
Statistical Analysis 1: Comparison: SpeediCath Catheter vs Conveen Uncoated; The analysis was done by comparing Kaplan-Meier estimates of the survival function of the two groups. The analysis was refined by a Cox proportional hazards regression model for survival data; Test type: Non-Inferiority or Equivalence — The additional explanatory variables were removed using backwards-elimination removing the least significant additional variable for each iteration, until the effect of all included additional variables was significant on α=0.05 significant level. The null-hypothesis of no catheter difference was to be rejected on α=0.05 significant level; p = 0.0383, Kaplan-Meier — p-value is adjusted for the following explanatory variables: catheterization frequency, technique (clean/sterile), procedure (participant/nurse), setting (hospital/community) and demographic measures; Hazard Ratio (HR) = 1.502, 95% CI 2-sided [1.022 to 2.207]

2. Secondary Outcome: UTIs With Bacteriuria >=100 Colony Forming Units (CFU)/ml
Description: UTIs with bacteriuria >=100 Colony Forming Units (CFU)/ml. Descriptive analysis
Time Frame: 4-6 months
Population: Descriptive only
Measure: Number; unit: UTI
Arm/Group | SpeediCath Catheter | Conveen Uncoated
Number analyzed (Participants) | 105 | 114
UTI | 101 | 151

3. Secondary Outcome: Nurse Evaluation of Catheters - Overall Satisfaction
Description: Evaluation score on an 11-point scale from 0-10 (0 being lowest satisfaction)
Time Frame: 4-6 months
Population: Analysis were done on evaluations of the ITT-population. Evaluations were made at discharge from hospital. Since some participants discontinued the study prior to discharge and since some did not fill in the evaluation form, the total number of evaluations (132) do not add up to the total of the ITT population (219)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | SpeediCath | Conveen Uncoated
Number analyzed (Participants) | 59 | 73
scores on a scale | 8.1 (2.3) | 8.3 (2.0)
Statistical Analysis 1: Comparison: SpeediCath vs Conveen Uncoated; Test type: Non-Inferiority or Equivalence — ANOVA analysis. Limit of significant difference <0.05; p = 0.7670, ANOVA — baseline characteristics were used as covariates, catheterization procedure (participant or caregiver) as well as technique (sterile or clean). Backward elimination was used

4. Secondary Outcome: Patient or Caregiver's Evaluation of Catheters - Overall Satisfaction
Description: Evaluation score on an 11-point scale from 0-10 (0 being lowest satisfaction)
Time Frame: 4-6 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | SpeediCath | Conveen Uncoated
Number analyzed (Participants) | 44 | 61
scores on a scale | 9.3 (1.4) | 8.6 (1.3)
Statistical Analysis 1: Comparison: SpeediCath vs Conveen Uncoated; Test type: Non-Inferiority or Equivalence — ANOVA. Level of significant difference <0.05; p = 0.0074, ANOVA — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Nurse Time Spent on Catheterization Procedure
Time Frame: 4-6 months
Population: ITT-population
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | SpeediCath | Conveen Uncoated
Number analyzed (Participants) | 38 | 53
seconds | 337 (44) | 278 (25)

6. Secondary Outcome: Device-related or Possibly Device-related AEs
Time Frame: 4-6 months
Measure: Number; unit: Events
Arm/Group | SpeediCath | Conveen Uncoated
Number analyzed (Participants) | 105 | 114
Events | 16 | 14

7. Secondary Outcome: Number of Participants With One or More Urinary Tract Infection
Time Frame: 4-6 months
Measure: Number; unit: participants
Arm/Group | SpeediCath | Conveen Uncoated
Number analyzed (Participants) | 105 | 114
participants | 47 | 82

ADVERSE EVENTS:
Arm/Group | SpeediCath | Conveen Uncoated
Serious Adverse Events (participants affected / at risk) | 5/105 | 6/114
Other Adverse Events (participants affected / at risk) | 16/105 | 14/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SpeediCath (N=105) | Conveen Uncoated (N=114)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 3 (3)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
subdural hematoma (General disorders) | 1 (1) | 0 (0) — not device-related
deep vein thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
urosepsis (Renal and urinary disorders) | 0 (0) | 1 (1)
perforated bladder/cystitis/decreased oxygen saturation (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SpeediCath (N=105) | Conveen Uncoated (N=114)
renal and urinary disorders (Renal and urinary disorders) | 16 (16) | 13 (13)
reproductive system and breast disorders (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less